CLINICAL TRIAL: NCT02157428
Title: Effect of Flumazenil on Recovery From General Anesthesia With Isoflurane: a Randomized Controlled Trial
Brief Title: Effect of Flumazenil on Recovery From General Anesthesia With Isoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Domingos Dias Cicarelli, MD, PhD, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 984/10
Record Dates: First submitted 2014-06-01; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Adverse Effect of Other General Anesthetics
MeSH Terms: interventions — Flumazenil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline (Placebo Comparator): patients received 20 ml of saline during 1 minute, after end of surgery.
  Interventions: Drug: saline
- flumazenil (Active Comparator): patients received 1 mg of flumazenil, after end of surgery
  Interventions: Drug: Flumazenil

INTERVENTIONS:
Drug: Flumazenil
  Arms: flumazenil
Drug: saline
  Arms: saline

SUMMARY:
Background and objectives: The inhalational anesthetic isoflurane is widely used in general anesthetics. Its mechanism of action involves interaction with the receptor of gamma-amino butyric acid (GABA), which is also the binding site for benzodiazepines. Flumazenil, benzodiazepine antagonist, reverses the effects of these drugs in GABA receptors and could therefore also reverse the effect of isoflurane. In anesthesia practice, extubation and early anesthetic recovery reduce morbidity and incidence of complications. The objective of this trial is to determine whether the use of flumazenil may contribute to faster recovery from anesthesia. Methods: 40 patients scheduled to undergo general anesthesia with isoflurane were enrolled in this prospective, double-blind, randomized trial. Patients were randomized to receive, at the end of anesthesia, flumazenil or placebo as allocated into two groups. The anesthetic technique was standardized. The groups were compared concerning values of Cerebral State Index (CSI), heart rate, blood pressure and oxygen saturation from the application of flumazenil or placebo until 30 minutes after injection. Data regarding time to extubation, time to reach ten points in the Aldrete-Kroulic score (AK = 10) and Vigilance score (VS = 10) was also collected. ANOVA test was applied to analyze the results, considering p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to surgeries with general anesthesia,
* healthy or with minor diseases completely controlled by regular use of medications (ASA I or II according to the classification of physical state by the American Society of Anesthesiologists).

Exclusion Criteria:

* patients with past of chronic use of benzodiazepines and/or illicit drugs,
* seizures or panic disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Time of recovery from a general anesthesia isoflurane based | up to 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário USP, São Paulo, São Paulo, Brazil